CLINICAL TRIAL: NCT00003871
Title: Phase II Randomized Study of Vaccine Treatment of Advanced Prostate Cancer
Brief Title: PSA Vaccine Therapy in Treating Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067036; E-7897
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: fowlpox virus vaccine vector
Biological: recombinant vaccinia prostate-specific antigen vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of different regimens of PSA vaccines in treating patients who have advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effect of prime and boost strategies using recombinant fowlpox prostate specific antigen (PSA) vaccine and recombinant vaccinia PSA vaccine on biochemical PSA progression in patients with stage D0 prostate cancer who have completed local treatment. II. Assess the tolerability and toxicity of these prime and boost treatment regimens in these patients. III. Evaluate the effects of these prime and boost treatment regimens on cellular immunity in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to HLA-2 typing (positive vs negative vs unknown). Patients are randomized to one of three treatment arms. Arm I: Patients receive intramuscular fowlpox prostate specific antigen (PSA) vaccine at weeks 0, 6, 12, and 18. Arm II: Patients receive intramuscular fowlpox PSA vaccine at weeks 0, 6, and 12 and intradermal vaccinia PSA vaccine at week 18. Arm III: Patients receive intradermal vaccinia PSA vaccine at week 0 and intramuscular fowlpox PSA vaccine at weeks 6, 12, and 18. Patients are followed at week 24, then every 3 months until year 2, every 6 months until year 5, and annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients (20 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven prostate cancer limited to the prostate (including seminal vesicle and/or local lymph node involvement) with elevated PSA (greater than 2 ng/ml) following surgery or rising PSA following radiotherapy Negative bone scan and CT scan of abdomen and pelvis No PSA progression during chemotherapy, hormonal therapy (including steroids), or neoadjuvant or adjuvant androgen ablation therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 6 months Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT and SGPT no greater than 2 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: Not specified Pulmonary: Not specified Other: No active untreated infection No known infection with HIV No concurrent medical conditions that would prevent compliance No history or evidence of active eczema or psoriasis or other contraindications to vaccinia virus administration (i.e., allergy) No significant allergy or hypersensitivity to eggs No evidence of immunosuppression Must be able to avoid contact with high risk individuals (immunosuppressed patients, children under 3, pregnant women, or patients with a history of or active eczema or other exfoliative diseases) for 7-10 days after immunization (household contacts must not be high risk) Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 6 months since prior chemotherapy and recovered Endocrine therapy: See Disease Characteristics At least 6 months since prior hormonal therapy (including steroids) and recovered Radiotherapy: See Disease Characteristics At least 3 months since prior radiotherapy of prostate and recovered Surgery: See Disease Characteristics At least 3 months since prior prostate surgery and recovered Other: Prior vaccinia immunization required OR Patient recollection of immunization and appropriate vaccination site scar

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1999-09-24 (Actual); Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard L. Kaufman, MD, Study Chair — Albert Einstein College of Medicine
Locations (10):
- United States (10):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Kaufman HL, Wang W, Manola J, et al.: Phase II prime/boost vaccination using poxviruses expressing PSA in hormone dependent prostate cancer: follow-up clinical results from ECOG 7897. [Abstract] J Clin Oncol 23 (Suppl 16): A-4501, 378s, 2005.
- [Result] Kaufman HL, Wang W, Manola J, DiPaola RS, Ko YJ, Sweeney C, Whiteside TL, Schlom J, Wilding G, Weiner LM. Phase II randomized study of vaccine treatment of advanced prostate cancer (E7897): a trial of the Eastern Cooperative Oncology Group. J Clin Oncol. 2004 Jun 1;22(11):2122-32. doi: 10.1200/JCO.2004.08.083. PMID 15169798
- [Result] Kaufman HL, Wang W, Manola J, et al.: Prime/boost vaccination using poxviruses expressing PSA in D0 prostate cancer: preliminary results of ECOG 7897, a randomized phase II clinical trial. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-12, 2002.